CLINICAL TRIAL: NCT07345494
Title: A Global Pregnancy Registry to Assess Maternal, Fetal, and Infant Outcomes Following Exposure to YORVIPATH® (Palopegteriparatide) During Pregnancy and Breastfeeding
Status: Not yet recruiting | Type: Observational
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ASND0043
Record Dates: First submitted 2025-11-24; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palopegteriparatide: Pregnant women exposed to palopegteriparatide during pregnancy
  Interventions: Drug: Palopegteriparatide

INTERVENTIONS:
Drug: Palopegteriparatide — Palopegteriparatide prescribed as per normal clinical practice

SUMMARY:
The purpose of this registry study is to collect both prospective and retrospective data in women exposed to palopegteriparatide during pregnancy to assess risk of pregnancy and maternal complications, and adverse effects on the developing fetus, neonate, and infant and to assess infant outcomes through at least the first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 15 to 50 years
* Participants with exposure to at least one dose of YORVIPATH at any time within 15 days prior to conception and/or during pregnancy. The timeframe of 15 days prior to conception is calculated based on 5 times the YORVIPATH half life of ~ 60 hours
* Participants providing written informed consent, verbal consent, or eConsent (depending on country regulations) and a Medical Release of Information. For adolescents under the age of majority, verbal or written informed assent by the pregnant minor (where applicable) and verbal or written informed consent by the parent/legal guardian will be obtained.

Exclusion Criteria:

* Pregnancies in which only the male partner is exposed to at least one dose of YORVIPATH.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with exposure to at least one dose of YORVIPATH at any time within 15 days prior to conception or during pregnancy. Prospective and retrospective pregnancies may be reported.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2036-01 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
The number of fetuses as reported by HCP | 21 months
Pregnancy outcomes | 21 months
  * Live birth (preterm delivery, full-term delivery)
  * Spontaneous abortion
  * Pregnancy termination
  * Fetal death/stillbirth
  * Molar or ectopic pregnancy
Number of congenital malformations identified in the developing fetus, neonate, or infant | 21 months
Descriptive statistics of adverse events (AEs), including serious adverse events (SAEs) | 21 months
Number of hospitalizations including reasons for hospitalization | 21 months
Descriptive statistics of growth and development milestones as described by the Centers for Disease Control and Prevention (CDC 2021) or other accepted standard assessment | 21 months
Number of signs of hypocalcemia or hypercalcemia | 21 months
Descriptive statistics of infant developmental deficiency (CDC 2021) | 21 months
Descriptive statistics of postnatal growth deficiency or failure to thrive (FTT) | 21 months
Descriptive statistics of neonatal and infant mortality | 21 months
Maternal complications of pregnancy | 21 months
  Including but not limited to
  * Premature rupture of membranes (PROM)
  * Preterm PROM (PPROM)
  * Pre-eclampsia
  * Gestational hypertension
  * Eclampsia
  * Proteinuria
  * Gestational diabetes
  * Intrauterine growth restriction (IUGR)
  * Polyhydramnios
  * Preterm delivery
  * Measures of fetal growth deficiency (e.g., small for gestational age)
Other maternal events of interest | 21 months
  Number of
  * AEs, including SAEs
  * Events specific to hypoparathyroidism (e.g., hypercalcemia, hypocalcemia). Serum calcium concentrations at each trimester (if available) and at birth

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Ascendis Pharma A/S